CLINICAL TRIAL: NCT02565082
Title: Evaluation of the Hemostatic Potential in Sickle Cell Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Dr Anne Demulder, Responsible of the Hematology laboratory, Brugmann University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-Drepanocytose-Hemostatic
Record Dates: First submitted 2015-09-18; First posted 2015-10-01 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Sickle Cell Disease
Keywords: Hemostatic potential; Sickle cell disease; Thrombin generation test
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sickle cell disease (Experimental): This arm will include an approximate number of 50 sickle cell disease patients, homozygous and heterozygous.
  Interventions: Other: Blood sampling - sickle cell patients arm - stable condition; Other: Blood sampling - sickle cell patients arm- exsanguinotransfusion needed; Other: Blood sampling - sickle cell patients arm - vaso-occlusive crisis.
- Control (Other): This arm will include an approximate number of 30 healthy volunteers.
  Interventions: Other: Blood sampling - healthy volunteers

INTERVENTIONS:
Other: Blood sampling - healthy volunteers — Four citrate blood sampling tubes (blue cap, 2.7ml) will be taken only once.
  Arms: Control
Other: Blood sampling - sickle cell patients arm - stable condition — Four citrate blood sampling tubes (blue cap, 2.7ml) will be taken only once.
  Arms: Sickle cell disease
Other: Blood sampling - sickle cell patients arm- exsanguinotransfusion needed — Four citrate blood sampling tubes (blue cap, 2.7ml) will be taken only once, before and after the exsanguinotransfusion.
  Arms: Sickle cell disease
Other: Blood sampling - sickle cell patients arm - vaso-occlusive crisis. — Four citrate blood sampling tubes (blue cap, 2.7ml) will be taken only once.
  Arms: Sickle cell disease

SUMMARY:
Sickle cell disease is a genetic disorder caused by a point mutation on the amino acid sequence of the β chain of hemoglobin.

The most expressive and most frequent complication of the disease is vaso-occlusive crisis, dominated by a painful syndrome. In addition to vaso-occlusive crises, many more chronic biological disturbances are observed in sickle cell patients.Sickle cell disease is considered nowadays as a hypercoagulable state.

However, the approach used so far to the measure of clotting in sickle cell disease was segmented in the sense that the various components of the hemostatic balance were studied separately.The thrombin generation test is a functional test which explores the coagulation globally, integrating both pro players that anticoagulants actors in the system. The investigators already used this test to demonstrate that the hemostatic potential was high in a cohort of affected children compared to control children of the same age.

This test will be used to characterize the hemostatic potential of adult sickle cell patients followed at the CHU Brugmann Hospital.

DETAILED DESCRIPTION:
Sickle cell disease is a genetic disorder caused by a point mutation on the amino acid sequence of the β chain of hemoglobin. This is the most common genetic disease in the world. The majority of patients are in Sub-Saharan Africa; however, the increase in migratory movements of populations helps to move patients out of the initial zones of the disease.

According to recent data, about 400 patients would be followed in the Belgian hospitals, and about 1 in 1500 newborns in Belgium would be a major carrier of hemoglobinopathies. The most expressive and most frequent complication of the disease is vaso-occlusive crisis, dominated by a painful syndrome. In addition to vaso-occlusive crises, many more chronic biological disturbances are observed in sickle cell patients. Their contribution to the course of the disease is becoming increasingly stressing. Among them are intravascular hemolysis, hyper-adhesion of blood cells to vascular endothelium, inflammation, oxidative stress, vasculopathy and bleeding disorders.

Sickle cell disease is considered nowadays as a hypercoagulable state. Indeed, sickle cell patients have a high risk of non-hemorrhagic stroke, thrombosis in the pulmonary arteries and deep vein thrombosis that are otherwise associated with mortality and high morbidity. Many anomalies at various levels in the hemostatic system demonstrate coagulation activation even in clinically stable condition.

However, the approach used so far to the measure of clotting in sickle cell disease was segmented in the sense that the various components of the hemostatic balance were studied separately. This scale is complex, this approach difficult to give a comprehensive and integrated picture of the various disturbances in the system. The thrombin generation test is a functional test which explores the coagulation globally, integrating both pro players that anticoagulants actors in the system. The investigators have used this test to demonstrate that the hemostatic potential was high in a cohort of affected children compared to control children of the same age. In this cohort high hemostatic potential was related to the rate of circulating microparticles and intravascular hemolysis rate. Studies are underway to look for correlations between the hemostatic potential and clinical complications in this pediatric cohort.

The use of thrombin generation test for the study of hemostasis in adult patients with sickle cell disease, and the contribution of coagulation disorders with the occurrence of complications of the disease remain little known. The investigators will therefore:

* Characterize the hemostatic potential of adult sickle cell patients followed at the CHU Brugmann
* Search for links between the hemostatic potential and other biological phenomena observed during the disease (intravascular hemolysis, microparticles, vasculopathy, inflammation)
* Search for correlations with clinical complications
* Evaluate the effect of treatment (including exchange transfusions) on the hemostatic potential.

ELIGIBILITY:
Inclusion Criteria:

- Sickle cell disease group: Sickle cell disease patients aged over 18 years

- Healthy volunteers group: Healthy volunteers, age matching with the sickle cell disease group

Exclusion Criteria:

- Sickle cell disease group: Pregnant women, dialysis patients, patients with an hepatic impairment, patients under treatments that can interfere with coagulation

- Healthy volunteers group: Pregnant women, known chronical disease, acute inflammatory syndrome, hemostasis disorder, abnormal complete blood count

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Coagulation markers | sickle cell patients - stable condition - at upcoming hospital routine follow-up, within maximum two years time
  The following coagulation markers will be assessed in the blood samples: thrombin and thrombomodulin, protein C, protein S, antithrombin, D-dimer, factor VIII, TFPI (physiological inhibitor of the extrinsic pathway of coagulation). This will be measured only once for each patient, for this health status.
Coagulation markers | sickle cell patients - if exsanguinotransfusion needed - immediately prior exsanguinotransfusion, within maximum two years time
  The following coagulation markers will be assessed in the blood samples:thrombin and thrombomodulin, protein C, protein S, antithrombin, D-dimer, factor VIII, TFPI (physiological inhibitor of the extrinsic pathway of coagulation). This will be measured only once for each patient, for this health status.
Coagulation markers | sickle cell patients - if exsanguinotransfusion needed - immediately after exsanguinotransfusion, within maximum two years time
  The following coagulation markers will be assessed in the blood samples:thrombin and thrombomodulin, protein C, protein S, antithrombin, D-dimer, factor VIII, TFPI (physiological inhibitor of the extrinsic pathway of coagulation). This will be measured only once for each patient, for this health status.
Coagulation markers | sickle cell patients - if vaso-occlusive crisis - during the vaso-occlusive crisis, within maximum two years time
  The following coagulation markers will be assessed in the blood samples:thrombin and thrombomodulin, protein C, protein S, antithrombin, D-dimer, factor VIII, TFPI (physiological inhibitor of the extrinsic pathway of coagulation). This will be measured only once for each patient, for this health status.
Coagulation markers | healthy volunteers: after informed consent signature, within maximum two years time
  The following markers will be assessed in the blood samples:thrombin and thrombomodulin, protein C, protein S, antithrombin, D-dimer, factor VIII, TFPI (physiological inhibitor of the extrinsic pathway of coagulation). This will be measured only once for each volunteer.
Hemolysis markers | sickle cell patients - stable condition - at upcoming hospital routine follow-up, within maximum two years time
  Will be measured in the blood samples by the following markers:plasmatic hemoglobin level and the lactate dehydrogenase level.This will be measured only once for each patient, for this health status.
Hemolysis markers | sickle cell patients - if exsanguinotransfusion needed - immediately prior exsanguinotransfusion, within maximum two years time
  Will be measured in the blood samples by the following markers:plasmatic hemoglobin level and the lactate dehydrogenase level.This will be measured only once for each patient, for this health status.
Hemolysis markers | sickle cell patients - if exsanguinotransfusion needed - immediately after exsanguinotransfusion, within maximum two years time
  Will be measured in the blood samples by the following markers:plasmatic hemoglobin level and the lactate dehydrogenase level.This will be measured only once for each patient, for this health status.
Hemolysis markers | sickle cell patients - if vaso-occlusive crisis - during the vaso-occlusive crisis, within maximum two years time
  Will be measured in the blood samples by the following markers:plasmatic hemoglobin level and the lactate dehydrogenase level.This will be measured only once for each patient, for this health status.
Hemolysis markers | healthy volunteers: after informed consent signature, within maximum two years time
  Will be measured in the blood samples by the following markers:plasmatic hemoglobin level and the lactate dehydrogenase level.This will be measured only once for each volunteer.
Microparticles level | sickle cell patients - stable condition - at upcoming hospital routine follow-up, within maximum two years time
  Will be measured in the blood samples both by a capture method (Zymuphen) and FACS.This will be measured only once for each patient, for this health status.
Microparticles level | sickle cell patients -if exsanguinotransfusion - immediately prior exsanguinotransfusion, within maximum two years time
  Will be measured in the blood samples both by a capture method (Zymuphen) and FACS. This will be measured only once for each patient, for this health status.
Microparticles level | sickle cell patients - if exsanguinotransfusion needed - immediately after exsanguinotransfusion, within maximum two years time
  Will be measured in the blood samples both by a capture method (Zymuphen) and FACS.This will be measured only once for each patient, for this health status.
Microparticles level | sickle cell patients - if vaso-occlusive crisis - during the vaso-occlusive crisis, within maximum two years time
  Will be measured both by a capture method (Zymuphen) and FACS.This will be measured only once for each patient, for this health status.
Microparticles level | healthy volunteers: after informed consent signature, within maximum two years time
  Will be measured in the blood samples both by a capture method (Zymuphen) and FACS. This will be measured only once for each patient, for this health status.
Inflammatory markers | sickle cell patients - stable condition - at upcoming hospital routine follow-up, within maximum two years time
  The following markers will be assessed in the blood samples: inflammatory cytokines, TNF, usCRP and interleukines. This will be measured only once for each patient, for this health status.
Inflammatory markers | sickle cell patients - if exsanguinotransfusion needed - immediately prior exsanguinotransfusion, within maximum two years time
  The following markers will be assessed in the blood samples: inflammatory cytokines, TNF, usCRP and interleukines. This will be measured only once for each patient, for this health status.
Inflammatory markers | sickle cell patients - if exsanguinotransfusion needed - immediately after exsanguinotransfusion, within maximum two years time
  The following markers will be assessed in the blood samples: inflammatory cytokines, TNF, usCRP and interleukines. This will be measured only once for each patient, for this health status.
Inflammatory markers | sickle cell patients - if vaso-occlusive crisis - during the vaso-occlusive crisis, within maximum two years time
  The following markers will be assessed in the blood samples: inflammatory cytokines, TNF, usCRP and interleukines. This will be measured only once for each patient, for this health status.
Inflammatory markers | healthy volunteers - after informed consent signature, within maximum two years time
  The following markers will be assessed in the blood samples: inflammatory cytokines, TNF, usCRP and interleukines. This will be measured only once for each volunteer.
Vascular markers | sickle cell patients - stable condition - at upcoming hospital routine follow-up, within maximum two years time
  The following markers will be assessed in the blood samples: soluble thrombomodulin, von Willebrand factor, vascular endothelial growth factor, protein C endothelial factor. This will be measured only once for each patient, for this health status
Vascular markers | sickle cell patients - if exsanguinotransfusion needed - immediately prior exsanguinotransfusion, within maximum two years time
  The following markers will be assessed in the blood samples: soluble thrombomodulin, von Willebrand factor, vascular endothelial growth factor, protein C endothelial factor. This will be measured only once for each patient, for this health status
Vascular markers | sickle cell patients - if exsanguinotransfusion needed - immediately after exsanguinotransfusion, within maximum two years time
  The following markers will be assessed in the blood samples: soluble thrombomodulin, von Willebrand factor, vascular endothelial growth factor, protein C endothelial factor. This will be measured only once for each patient, for this health status
Vascular markers | healthy volunteers - after informed consent signature, within maximum two years time
  The following markers will be assessed in the blood samples: soluble thrombomodulin, von Willebrand factor, vascular endothelial growth factor, protein C endothelial factor. This will be measured only once for each volunteer.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Demulder, MD, Principal Investigator — CHU Brugmann; Bhavna Mahadeb, Principal Investigator — St Pierre Hospital
Locations (1):
- CHU Brugmann Hospital, Brussels, Belgium

REFERENCES:
- [Background] Le PQ, Ferster A, Cotton F, Vertongen F, Vermylen C, Vanderfaeillie A, Dedeken L, Heijmans C, Ketelslegers O, Dresse MF, Gulbis B. Sickle cell disease from Africa to Belgium, from neonatal screening to clinical management. Med Trop (Mars). 2010 Dec;70(5-6):467-70. PMID 21516988
- [Background] Rees DC, Williams TN, Gladwin MT. Sickle-cell disease. Lancet. 2010 Dec 11;376(9757):2018-31. doi: 10.1016/S0140-6736(10)61029-X. Epub 2010 Dec 3. PMID 21131035
- [Background] Ataga KI, Key NS. Hypercoagulability in sickle cell disease: new approaches to an old problem. Hematology Am Soc Hematol Educ Program. 2007:91-6. doi: 10.1182/asheducation-2007.1.91. PMID 18024615
- [Background] De Franceschi L, Cappellini MD, Olivieri O. Thrombosis and sickle cell disease. Semin Thromb Hemost. 2011 Apr;37(3):226-36. doi: 10.1055/s-0031-1273087. Epub 2011 Mar 31. PMID 21455857
- [Background] Manci EA, Culberson DE, Yang YM, Gardner TM, Powell R, Haynes J Jr, Shah AK, Mankad VN; Investigators of the Cooperative Study of Sickle Cell Disease. Causes of death in sickle cell disease: an autopsy study. Br J Haematol. 2003 Oct;123(2):359-65. doi: 10.1046/j.1365-2141.2003.04594.x. PMID 14531921
- [Background] Hemker HC, Giesen P, Al Dieri R, Regnault V, de Smedt E, Wagenvoord R, Lecompte T, Beguin S. Calibrated automated thrombin generation measurement in clotting plasma. Pathophysiol Haemost Thromb. 2003;33(1):4-15. doi: 10.1159/000071636. PMID 12853707
- [Background] Noubouossie DF, Le PQ, Corazza F, Debaugnies F, Rozen L, Ferster A, Demulder A. Thrombin generation reveals high procoagulant potential in the plasma of sickle cell disease children. Am J Hematol. 2012 Feb;87(2):145-9. doi: 10.1002/ajh.22206. Epub 2011 Nov 4. PMID 22052675
- [Background] Noubouossie DC, Le PQ, Rozen L, Debaugnies F, Ferster A, Demulder A. Evaluation of the procoagulant activity of endogenous phospholipids in the platelet-free plasma of children with sickle cell disease using functional assays. Thromb Res. 2012 Aug;130(2):259-64. doi: 10.1016/j.thromres.2011.10.016. Epub 2011 Nov 12. PMID 22079446